CLINICAL TRIAL: NCT03889847
Title: Comparison of Fiberoptic Bronchoscopic Intubation Between Silicone and Polyvinylchloride Double Lumen Tube.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, DAE HEE KIM, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AJIRB-DEV-THE-18-44-
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Intubation;Difficult
Keywords: Fiberoptic intubation; double lumen tube

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- silicone DLT (Experimental): Fibreoptic intubation with silicone double lumen tube
  Interventions: Device: Fibreoptic intubation with silicone double lumen tube
- PVC DLT (Experimental): Fibreoptic intubation with PVC double lumen tube
  Interventions: Device: Fibreoptic intubation with PVC double lumen tube

INTERVENTIONS:
Device: Fibreoptic intubation with silicone double lumen tube — Fibreoptic intubation with silicone double lumen tube
  Arms: silicone DLT
Device: Fibreoptic intubation with PVC double lumen tube — Fibreoptic intubation with PVC double lumen tube
  Arms: PVC DLT

SUMMARY:
One lung ventilation (OLV) is required during thoracic procedure such as lung and esophagus surgery, and carried out by double lumen tube(DLT). Direct insertion of DLT over a fibreoptic bronchoscope (FOB) is considered more difficult and traumatic than that of a single-lumen tube. Recently, One recent simulation study demonstrated that a soft silicone DLT with a flexible, wire-reinforced bronchial tip (Fuji-Phycon tube) may shorten the time to intubation via tube exchange when compared with less compliant, polyvinyochloride(PVC) DLTs such as the Shilly or Rusch DLT. HumanBroncho® (Insung Medical, Seoul, Korea) is a new silicone DLT with a soft, flexible, non-bevelled, wire-reinforced tip. The oval shape, obtuse angle, and short lateral internal diameter of the bronchial lumen and its flexibility may allow for advancement to the trachea over the FOB easier than the Shilly tube.

In the present study, The investigators aimed to test the hypothesis that the silicone DLT would be easier than PVC DLT with regard to railroading grade over an FOB. Investigators further aimed to compare the intubation time over the FOB between the silicone DLT and PVC DLT.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracic surgery and one lung ventilation American Society of Anesthesiologist physical status 1,2

Exclusion Criteria:

* abnormal upper airway, gastrointestinal disease, risk of aspiration, BMI > 35

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
railroading grade | an average of 2 minutes
  grade of ease of railroading over fibreoptic bronchoscope.
  1. no difficulty passing the tube
  2. obstruction while passing the tube, relieved by withdrawal and 90 degree counter-clockwise rotation(2-1) or more than 90 degree rotation(2-2)
  3. obstruction necessitating more than one manipulation or external laryngeal manipulation
  4. direct laryngoscope was required

SECONDARY OUTCOMES:
insertion time | an average of 2 minutes
  time from insertion of FOB into mouth to tube placement into trachea and left main bronchus
number of patients with trauma around glottis, observed by FOB | an average of 2minutes
  glottic trauma observation through FOB outside the tube
number of patients with tube repositioning during the surgery | an average of 3.5 hours
  count of tube repositioning with FOB during the surgery
number of patients with complication of hoarseness, sore throat, and swallowing difficulty | an average of 30 minutes
  hoarseness, sore throat, swallowing difficulty in post-anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hee Kim, M.D., Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou universiry hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No